CLINICAL TRIAL: NCT07227818
Title: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Assess the Efficacy of NBI-1117568 in Preventing Relapse of the Symptoms of Schizophrenia and to Assess the Safety and Tolerability of NBI-1117568 in Adults With Schizophrenia
Brief Title: Efficacy of NBI-1117568 in Preventing Relapse in Adults With Schizophrenia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1117568-SCZ3031
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NBI-1117568
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The initial Open-label Stabilization Period is open-label and non-randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-1117568 (Experimental): All participants will receive NBI-1117568 during the Open-label Stabilization Period, then will be randomized to receive NBI-1117568 during the Double-blind Treatment Period.
  Interventions: Drug: NBI-1117568
- Placebo (Placebo Comparator): All participants will receive NBI-1117568 during the Open-label Stabilization Period, then will be randomized to receive placebo matching NBI-1117568 during the Double-blind Treatment Period.
  Interventions: Drug: NBI-1117568; Drug: Placebo

INTERVENTIONS:
Drug: NBI-1117568 — Oral capsules
Drug: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate NBI-1117568 compared with placebo in delaying relapse of symptoms of schizophrenia in adults who have a stable response after open-label treatment with NBI-1117568.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria.
* Participant had the initial diagnosis of schizophrenia ≥1 year before screening.
* Participant has had a positive response to ≥1 antipsychotic therapy (other than clozapine) at a therapeutic dose.

Key Exclusion Criteria:

* Participant has an unstable or poorly controlled medical condition or chronic disease (including history of neurological [including dementing illness, myasthenia gravis], hepatic, renal, cardiovascular, gastrointestinal, pulmonary, autoimmune, or endocrine disease that may affect study participation or results) or malignancy within 30 days before Day 1.
* Participant has any laboratory abnormalities suggestive of clinically significant, poorly managed, or unmanaged undiagnosed disease.
* Participant has a history of clozapine treatment for treatment-resistant psychosis.
* Participant has a history of a stay in a psychiatric inpatient facility for ≥30 consecutive days (other than for purely social reasons or due to participation in a different clinical trial) during the 90 days before screening.
* Participant has initiated or increased intensity of nonpharmacological psychosocial therapeutic treatment within 3 weeks before screening or is expected to change throughout the length of the study.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Time From Randomization to Relapse | Up to approximately 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences